CLINICAL TRIAL: NCT00612391
Title: A Randomized Clinical Trail Comparing a Lateral Minimally Invasive Approach and the Traditional Anterior Approach for Plating of Proximal Humerus Fractures
Brief Title: Lateral Mini Approach vs Anterior Approach for Plating of Proximal Humerus Fracture
Acronym: HURA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Dominique Rouleau, Orthopaedic surgeon, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HURA1
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Closed Fracture Proximal Humerus, Neck
Keywords: humerus fracture
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lateral, Minimally Invasive Approach (Experimental): Lateral, Minimally Invasive Approach in GT fractures treated operatively (plates and screws)
  Interventions: Procedure: Lateral minimally invasive approach (plate fixation)
- Deltopectoral approach: (Active Comparator): Deltopectoral approach for GT fracture treated operatively
  Interventions: Procedure: Deltopectoral approach (plate fixation)

INTERVENTIONS:
Procedure: Lateral minimally invasive approach (plate fixation) — A longitudinally oriented, 4-cm incision will be made laterally starting at the acromion. The deltoid will be split proximally at the most strategic location (vis-à-vis the fracture), and after the deltoid is bluntly elevated from the humerus more distally the axillary nerve will be identified by digital palpation. The nerve is easily identified posteriorly as it emerges from the quadrilateral space. With a finger maintained on the nerve for protection, the plate will be inserted onto the lateral side of the proximal humerus and fixed according to the described technique. A second, 2-cm longitudinal incision will then be made further distally for diaphyseal screw placement. This incision is well distal to the course of the axillary nerve.
  Arms: Lateral, Minimally Invasive Approach
Procedure: Deltopectoral approach (plate fixation) — Anterior, Delto-Pectoral Approach - A 10-cm incision will be made over the deltopectoral groove, starting at the coracoid process proximally. As the clavipectoral fascia is incised, the cephalic vein will be identified and retracted laterally with the deltoid muscle. The pectoralis major as well as the conjoint tendon will be retracted medially, and the long head of the biceps tendon will be identified and used as a guide for achieving an anatomic reduction of the different fracture parts. Next, internally rotating the humerus will allow access to the lateral side of the proximal humerus, on which the plate will then be fixed according to the described technique.
  Arms: Deltopectoral approach:

SUMMARY:
A prospective randomized clinical trial is proposed to compare the plate fixation of proximal humerus fractures using a minimally invasive lateral approach and the traditional anterior approach.Forty five patients will be assigned to each approach (total of 90 patients) and will be assessed 7 times over a two-year period. The trial's primary objectives will be to demonstrate the efficacy of the plating technique in terms of speed of recuperation of function. The Quick DASH will be used for evaluation of function.The study will also examine secondary end-points of pain, range of motion, esthetic satisfaction and radiographic outcome, as assessed by the components of the Constant Score3,4, SF-12V2 Questionnaire, and Patient Scare Assessment Scale Questionnaire. Furthermore, the assessment of safety will be based on the rates of all reported complications and adverse events at 2 years

ELIGIBILITY:
Inclusion Criteria:

1. Humeral surgical neck fracture, Neer II valgus-type Neer III
2. Patient willing to participate in the study
3. Patient available for follow-up through at least two years
4. Patient with acceptable preoperative medical clearance and free of, or treated for, medical conditions that would pose excessive operative risk
5. Patient fluent in French and/or English and able to understand his/her role in the study

Exclusion Criteria:

1. Inflammatory arthritis
2. Prior shoulder pathology
3. Active local or systemic infection
4. Neurologic or musculoskeletal disease that may adversely affect mobility
5. Participation in any other pharmaceutical, biologic or medical-device clinical investigation
6. Severe documented psychiatric disease
7. Severe ipsilateral elbow or wrist disease
8. Fracture resistant to reduction attempts through the minimally invasive lateral approach

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-11; Primary Completion 2019-07 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Quick DASH | 3, 6, and 12 weeks, and at 6, 12, 18 and 24 months.

SECONDARY OUTCOMES:
SF-12V2 Questionnaire Constant Shoulder Score The Patient Scar Assessment Scale Complication rate | 3, 6, and 12 weeks, and at 6, 12, 18 and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique M Rouleau, MD, Principal Investigator — Hopital Sacré-Coeur
Locations (1):
- Hopital Sacré-Coeur, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196